CLINICAL TRIAL: NCT06547671
Title: Evaluation of the Effectiveness of a Comfort-sensory Room in the Control of Agitation in a Functional Mental Health Rehabilitation Area
Brief Title: Efficacy of a Sensory Comfort Room in Agitation Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioaraba Health Research Institute (Network)
Responsible Party: Principal Investigator, Maria Olárizu Olalde Ortiz, Nurse in Araba University Hospital, Bioaraba Health Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGITCONF2024
Record Dates: First submitted 2024-07-08; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Mental Disorders, Severe
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Not randomized clinical trial in parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comfort room (Experimental): Use of the sensory comfort room located in the unit itself, decorated in soft and relaxing tones with motifs inspired by nature. It has relaxation sofas, rocking chair, aromatherapy, chromotherapy, projector, music of the user's choice, weighted blanket mats, balls of various sizes......... to teach people admitted to the area alternatives to cope and control anxiety and prevent the escalation of agitation, as well as to guide them in strategies to help them relax.
  In addition, as usual clinical practice, both before and after the intervention, verbal de-escalation techniques will be used, for which the professionals in the area have been trained with a verbal de-escalation course specifically for working in the area.
  The intervention is not unique but in several uses of the sensory comfort room in each patient. The intervention will last approximately 30 minutes and can be used several times during the day. Furthermore, patients received the same follow up than the control group.
  Interventions: Other: Employment of a confort room to help in anxiety and agitation moments.
- Usual clinical practice (No Intervention): Follow up of patients, in the same way as in routine clinical practice.

INTERVENTIONS:
Other: Employment of a confort room to help in anxiety and agitation moments. — Use of the sensory comfort room located in the unit itself, decorated in soft and relaxing tones with motifs inspired by nature. It has relaxation sofas, rocking chair, aromatherapy, chromotherapy, projector, music of the user's choice, weighted blanket mats, balls of various sizes......... to teach people admitted to the area alternatives to cope and control anxiety and prevent the escalation of agitation, as well as to guide them in strategies to help them relax.
  Arms: Comfort room

SUMMARY:
In the initial approach of the study, it was considered that the comfort room would be used by all patients with GCT treated in the Functional Rehabilitation Area 1 (ARF 1) of the Álava Psychiatric Hospital. However, with the onset of the covid-19 pandemic, the service itself decided to separate the patients into two units, in order to reduce positive contacts. Consequently, the use of the comfort room will only be available for one of the two units, which will be considered as the intervention group, while the other unit will be considered as the control group. It is also important to note that the patients in the intervention group unit have a more severe mental state than those in the control group. The control group are older and more psychopathologically stable patients. So already from the initial moment of the study they are two populations with different characteristics.

Main Objective:

To determine the effectiveness of the use of a sensory comfort room in the functional rehabilitation area 1 of the HPA. It would be considered effective if mechanical restraints decrease by 5% in the intervention group with respect to the previous year.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to functional rehabilitation area 1 presenting with questionable, mild or moderate Agitation (score less than or equal to 20 on the PEC scale) or at the patient's request.
* To have freely accepted to participate in the intervention and to have signed the informed consent. An information sheet will also be given to the patient and an information sheet to the tutor (APPENDIXES 1 and 2). Experts in easy reading are consulted to adapt this document.

Exclusion criteria:

* Severe and extremely severe agitation (score greater than or equal to 21 on the PEC scale). Immediate previous physical aggression.
* Declination of the signature of informed consent.
* Any participant who does not comply with the rules of use of the room will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Number of mechanical restraints | Up to 24 months
  Mechanical restraint is understood as the extreme therapeutic intervention, through the application of immobilizing restrictive devices to limit a patient's freedom and, in turn, allows us to ensure their own safety and/or that of other

SECONDARY OUTCOMES:
Change in the agitation level | Through study completion, an average of 2 years
  Agitation Score in Positive and Negative Symptoms Scale, Excitement Component (PEC) It is a scale with five items: Tension; Uncooperativeness; Hostility; Poor impulse control; and Excitement. Each of these items is rated with the following scores: 1. Absent. 2. Minimal. 3. Mild. 4. Moderate. Moderately severe. 6. Severe. 7. Extreme.
  A higher score on the PEC scale indicates greater agitation. The classification of the level of agitation is as follows: Questionable (5-10 points), mild (11-15 points) Moderate (16-20 points) Moderately severe (20-25 points) Severe (26-30 points or Item "impulse control" > 4) Extremely severe (30-35 points).
  Whether or not the score on the PEC scale is lower before using the room and afterwards will be evaluated (15). It is considered that there is a decrease in the PEC scale if it is lower by one point. Before room use and afterwards.
Number of isolations | Up to 24 months
  Defined as the supervised confinement of a patient in a locked room alone for a period of time to protect the patient, or staff, from serious harm
Number of patients who need Rescue medication | Up to 24 months
  Rescue medication to overcome the crisis

OTHER OUTCOMES:
Patients satisfaction questionnaire with confort room | Through study completion, an average of 2 years
  Satisfaction and Proposals for room improvement, completed after each use
Professionals satisfaction questionaire with confort room | Through study completion, an average of 2 years
  About their experience with the employment of room, completed after each use
Age | At baseline
  Numerical variable
Sex | At baseline
  Male, famale
Cognitive level with mini-mental scale. | At baseline
  This is the most widely used brief cognitive test in Spain. It is mainly used to detect cognitive disorders associated with neurodegenerative diseases such as Alzheimer's disease. There are 2 versions of 30 and 35 points. The test has 5 items (orientation, fixation, concentration and calculation, memory, language and construction). Impairment is considered to be present when the score is less than 23 points
Age of mental disease evolution | At baseline
  Numerical variable
Diagnosis | At baseline
  According to the International Classification of Diseases

CONTACTS AND LOCATIONS:
Overall Officials: MARIA OLÁRIZU OLALDE, Principal Investigator — Basque Health Service
Locations (1):
- Araba University Hospital, Vitoria-Gasteiz, Alava, Spain